CLINICAL TRIAL: NCT06367855
Title: Efficacy and Safety of Preemptive Intravenous Dexamethasone in MIS-TLIF
Acronym: MIS-TLIF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Potsawat Surabotsopon (Other)
Responsible Party: Sponsor-Investigator, Potsawat Surabotsopon, MD, Thammasat University Hospital
Organization: Thammasat University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KSKC20222025
Record Dates: First submitted 2024-03-24; First posted 2024-04-16 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-04

CONDITIONS: Spinal Stenosis Lumbar; Disc Degeneration; Disc Disease; Fusion of Spine; Surgery
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone group (Active Comparator)
  Interventions: Drug: Dexamethasone
- Normal saline group (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — long-acting corticosteroid IV route
  Arms: Dexamethasone group
Drug: Normal saline — normal saline
  Arms: Normal saline group

SUMMARY:
Researchers are considering Dexamethasone as preemptive medication before minimally invasive spine fusion surgery to minimize postoperative back pain with minimal side effects, aiming to enhance the effectiveness of surgery and improve patient outcomes.

DETAILED DESCRIPTION:
Surgery for spine fusion through a minimally invasive technique called MIS-TLIF has become increasingly popular nowadays due to various reasons such as lower blood loss and reduced need for blood transfusions, less postoperative back pain, and shorter surgical duration compared to the traditional technique known as TLIF. However, even after MIS TLIF, patients still experience issues such as wound or back pain, which can affect their physical activity and increase the risk of infection. Prolonged hospital stays lead to resource wastage.

In the Enhanced Recovery After Surgery (ERAS) program for spine surgery, preoperative medication, including Acetaminophen, NSAIDs, and Gabapentinoids, is recommended to alleviate postoperative back pain. However, even after implementing ERAS, patients undergoing MIS TLIF still experience pain, suggesting that further pain reduction strategies are needed. The use of Dexamethasone as preemptive medication has shown promising results in various surgeries, with minimal side effects and a manageable cost. Dexamethasone, administered via injection, has a longer duration of action compared to other steroids, making it suitable for preemptive use.

The main objective is to study the effectiveness of using Dexamethasone via intravenous injection before minimally invasive spine fusion surgery, known as MIS-TLIF, in reducing postoperative back pain.

The secondary objectives are to compare the rate of morphine usage for pain management after surgery between two groups.

To compare the side effects and adverse reactions of the medication, such as nausea and vomiting, surgical site infection rates, and blood sugar levels post-surgery.

To compare the fusion rates of the spinal bones. To compare the length of hospital stays after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 50-80 years old.
* Undergoing MIS TLIF surgery at 1-2 spinal levels.

Exclusion Criteria:

* Previously undergone spine surgery.
* HbA1C greater than or equal to 7.5 mg%
* Allergic to all types of experimental medication.
* History of using systemic steroids.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
effectiveness of dexamethasone | 24 hours, 2 weeks, 6 weeks, 12 weeks post operative period
  postoperative VAS score at rest and motion for back pain

SECONDARY OUTCOMES:
Morphine consumption | 24 hours post operative period
  rate of morphine usage for pain management
Complication | 24 hours, 2 weeks, 6 weeks, 12 weeks post operative period
  To compare the side effects and adverse reactions of the medication, such as nausea and vomiting, surgical site infection rates, and blood sugar levels post-surgery
Fusion rate | 6months
  To compare the fusion rates of the spinal bones
Length of hospital stay | 1 year
  To compare the length of hospital stays after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat university hospital, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
data request can be submitted 1 year after publication and available up to 2 years
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: data request can be submitted 1 year after publication and available up to 2 years
Access Criteria: access to IPD can be requested to the first researcher's email as noted in this form

REFERENCES:
- [Background] Mobbs RJ, Phan K, Malham G, Seex K, Rao PJ. Lumbar interbody fusion: techniques, indications and comparison of interbody fusion options including PLIF, TLIF, MI-TLIF, OLIF/ATP, LLIF and ALIF. J Spine Surg. 2015 Dec;1(1):2-18. doi: 10.3978/j.issn.2414-469X.2015.10.05. PMID 27683674
- [Background] Goldstein CL, Macwan K, Sundararajan K, Rampersaud YR. Comparative outcomes of minimally invasive surgery for posterior lumbar fusion: a systematic review. Clin Orthop Relat Res. 2014 Jun;472(6):1727-37. doi: 10.1007/s11999-014-3465-5. PMID 24464507
- [Background] Lee MJ, Mok J, Patel P. Transforaminal Lumbar Interbody Fusion: Traditional Open Versus Minimally Invasive Techniques. J Am Acad Orthop Surg. 2018 Feb 15;26(4):124-131. doi: 10.5435/JAAOS-D-15-00756. PMID 29337717
- [Background] Debono B, Wainwright TW, Wang MY, Sigmundsson FG, Yang MMH, Smid-Nanninga H, Bonnal A, Le Huec JC, Fawcett WJ, Ljungqvist O, Lonjon G, de Boer HD. Consensus statement for perioperative care in lumbar spinal fusion: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Spine J. 2021 May;21(5):729-752. doi: 10.1016/j.spinee.2021.01.001. Epub 2021 Jan 12. PMID 33444664
- [Background] Salerno A, Hermann R. Efficacy and safety of steroid use for postoperative pain relief. Update and review of the medical literature. J Bone Joint Surg Am. 2006 Jun;88(6):1361-72. doi: 10.2106/JBJS.D.03018. PMID 16757774
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- [Background] Tammachote N, Kanitnate S. Intravenous Dexamethasone Injection Reduces Pain From 12 to 21 Hours After Total Knee Arthroplasty: A Double-Blind, Randomized, Placebo-Controlled Trial. J Arthroplasty. 2020 Feb;35(2):394-400. doi: 10.1016/j.arth.2019.09.002. Epub 2019 Sep 7. PMID 31587982
- [Background] Bednar DA, Wong A, Farrokhyar F, Paul J. Dexamethasone Perioperative Coanalgesia in Lumbar Spine Fusion: A Controlled Cohort Study of Efficacy and Safety. J Spinal Disord Tech. 2015 Aug;28(7):E422-6. doi: 10.1097/BSD.0b013e3182a1ddd3. PMID 26213843
- [Background] Jeyamohan SB, Kenning TJ, Petronis KA, Feustel PJ, Drazin D, DiRisio DJ. Effect of steroid use in anterior cervical discectomy and fusion: a randomized controlled trial. J Neurosurg Spine. 2015 Aug;23(2):137-43. doi: 10.3171/2014.12.SPINE14477. Epub 2015 May 1. PMID 25932600